CLINICAL TRIAL: NCT01881139
Title: Effects of Exercise Training on Cardiac Function and Lipid Metabolism in Mem 18-22 Year Old
Brief Title: Impact of Exercise Training on Cardiac Function in Man
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: No. 150 Central Hospital of the Chinese People Liberation Army (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 150CTSX002
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cardiovascular Disease
Keywords: Exercise; Lipid; Left ventricular; heart function
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental 1 (Experimental): men with exercise training for 3 months
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training

SUMMARY:
The purpose of this study is to monitor the impact of exercise training on cardiac functions and lipoprotein lipids.

DETAILED DESCRIPTION:
Exercise can increase the mass of left ventricle, which is also called athletic heart. Athletic heart is most frequently encountered as a pathological manifestation of cardiovascular disease, and the early determinants of athelitic remodeling in the general population are largely unknown. We will recruit 45 men aged 18-25 years who will run 5000 meters 2/day for 3 months. caridac function is examined by ECG and echocardiogram, blood pressure, lipoprotein, heart rate, body weight, cardiac troponin will be examined prior to exercise program and 3 months after exercise.

ELIGIBILITY:
Inclusion Criteria:

* men
* age 18-25 years
* body mass index (BMI) 18-25 kg/m2
* no regular exercise
* no tobacco use
* no current use of prescribed medications
* no self-report of acute of chronic diseases

Exclusion Criteria:

* conditions that do not meet the inclusion criteria listed.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change of cardiac function at baseline to exercise training for 3 months | baseline to 3 months

SECONDARY OUTCOMES:
change of lipoprotein at baseline to exercise training for 3 months | baseline to 3 months
change of heart rate at baseline to exercise training for 3 months | baseline to 3 months
Change of body weight at baseline to exercise training for 3 months | baseline to 3 months
change of cardiac troponin frome baseline to exercise training for 3 months | baselin to 3 months
Change of blood pressure from baseline to exercise training for 3 months | baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shenxu Wang, MD, Study Director — No. 150 Central Hospital of PLA
Locations (1):
- No. 150 Central hospital of Chinese People's Liberation Army, Luoyang, Henan, China